CLINICAL TRIAL: NCT01312155
Title: Assisted Intubation
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Thomas Hemmerling, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 10-338
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Intubation Conditions
Keywords: endotracheal; intubation; video; time
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing general anesthesia
  Interventions: Other: Intubation

INTERVENTIONS:
Other: Intubation — Intubation, endotracheal

SUMMARY:
The study investigates assisted intubation using a videolaryngoscope in anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Easy airway assessment

Exclusion Criteria:

* Difficult airway
* ASA 3

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia with endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Performance | 3 months
  Success rate in % of intubation: Number of patients where 'assisted intubation' was successful

SECONDARY OUTCOMES:
Time | 3 months
  Time to intubate: time in sec between insertion of scope into mouth and insertion of endotracheal tube through vocal cords

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hemmerling, MD, Principal Investigator — MUHC - McGill
Locations (1):
- MUHC, Montreal, Quebec, Canada